CLINICAL TRIAL: NCT02067442
Title: Prospective, Randomized, Double-blind, Placebo-Controlled Study to Compare the Effects of Intravenous Versus Oral Acetaminophen on Postoperative Clinical Outcomes After Ambulatory Lumbar Discectomy
Brief Title: Prospective, Randomized, Double Blind Study Comparing IV vs PO Acetaminophen in Patients Undergoing Lumbar Discectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 12D.685
Record Dates: First submitted 2014-01-17; First posted 2014-02-20 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Pain
Keywords: acetaminophen intravenous oral pain scores opioids
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral acetaminophen (Active Comparator): Patients in this arm of the study will receive oral acetaminophen and an IV placebo
  Interventions: Drug: oral acetaminophen
- intravenous acetaminophen (Active Comparator): Patients in this arm of the study will receive IV acetaminophen and an oral placebo
  Interventions: Drug: intravenous acetaminophen

INTERVENTIONS:
Drug: oral acetaminophen — 1000 milligrams given orally before surgery
  Other Names: Tylenol
  Arms: oral acetaminophen
Drug: intravenous acetaminophen — 1000 milligrams of intravenous acetaminophen given before surgery
  Other Names: Ofirmev
  Arms: intravenous acetaminophen

SUMMARY:
Both intravenous and oral acetaminophen have been shown to reduce post-operative pain scores when given preoperatively. This study investigates if there is a difference between the intravenous and the oral forms when given preoperatively to patients undergoing lumbar microdiscectomy. We hypothesize that the intravenous formulation does not improve pain scores or decrease opioid consumption during the first postoperative day compared to the oral formulation.

ELIGIBILITY:
Inclusion Criteria:

* Single level lumbar micro disk surgery
* Ages 18-65

Exclusion Criteria

* morbid obesity
* prior back surgery
* opioid tolerance
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain scores | Day of surgery
  Pain scores are measured using a visual analog scale with patient at rest and also with movement of the lower extremities at four separate times following surgery.

SECONDARY OUTCOMES:
Quantity of intraoperative and postoperative opioids administered. | Day of surgery
  All doses of opioids given on the day of surgery will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hopsital, Philadelphia, Pennsylvania, United States